CLINICAL TRIAL: NCT00352326
Title: Optimizing Assisted Communication Devices for Children With Motor Impairments Using a Model of Information Rate and Channel Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Terence Sanger, Associate Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FITTS PILOT
Record Dates: First submitted 2006-07-12; First posted 2006-07-14 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children (with dystonia and controls) (Experimental): Participants sat in a chair or their own wheelchair in front of a table whose surface height was adjusted at the midpoint between the hip and the Xiphoid process. They placed the hand that was not used for the task on their lap.
  An iPad® (Apple Inc, Cupertino, California) was located on the table in portrait mode in front of the participants at a distance that ranged between 40 and 55 cm. An adjustable metal bookstand supported the iPad® to allow the participants a comfortable screen view. The size of the screen was 19.5 × 14.6 cm. Custom software was developed for the experimental task (XCode 3.2 development environment, iOS 4.2 operating system; Apple Inc, Cupertino, California).
  Interventions: Device: reprogramming assisted communication device interface

INTERVENTIONS:
Device: reprogramming assisted communication device interface — The subjects were required to touch targets on the iPad® screen with the index finger of their preferred (less-affected) arm. The experimental task consisted of 180 targets divided in 4 blocks: 45 targets each block with a 1-minute interval between trials to avoid fatigue. Targets appeared at 1 of 9 different locations on the screen, and subjects moved their finger sequentially from one target to the next.

SUMMARY:
For children who depend on devices to communicate, the rate of communication is a primary determinant of success. For children with motor impairments, the rate of communication may be limited by inability to contact buttons or cells rapidly or accurately. It is therefore essential to know how to adjust the device interface in order to maximize each child's rate of communication. The optimal rate of communication is determined by the Channel Capacity, which is the maximum value of the Information Rate for all possible keyboard button or cell layouts for the communication device. We construct a mathematical model for the information rate based on the relationship between movement time and the number of buttons per screen, the size of the buttons, and the length of a sequence of buttons that must be pressed to communicate each word in the vocabulary. We measure the parameters of the model using a custom-programmed touch-screen interface.

ELIGIBILITY:
Inclusion Criteria:- Use of Dynavox ability to follow two-step commands impairment in arm function Exclusion Criteria:- increased risks of study

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2006-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence D. Sanger, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States